CLINICAL TRIAL: NCT06193265
Title: Management of Lumbar Discectomy by Endoscopy and Conventional Microscopic Discectomy
Acronym: ENDOLOMB
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: RGDS-2022-06-025
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Diskectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery under full endoscopy: A full endoscopic surgery will be performed on patienst with herniated disc
  Interventions: Procedure: Discectomy
- Conventional microscopic surgery: A conventional microscopic surgery will be performed on patienst with herniated disc
  Interventions: Procedure: Discectomy

INTERVENTIONS:
Procedure: Discectomy — Discectomy is total or more often partial intervertebral disc surgical removal

SUMMARY:
Currently, microscopic discectomy is performed as a minimally invasive surgery, thus reducing impact of so-called conventional "open" discectomies.

Although more technically demanding, discectomy with full endoscopy made possible a significant reduction of surgery invasive impact, thus making possible to broaden the field of endoscopic surgery indications.

This study is based on hypothesis that complete endoscopic discectomy offers several advantages over traditional microscopic discectomy, including a smaller skin incision and therefore fewer scars and less muscle damage, lower infection rate, less blood loss, less painful post-operative recovery and shorter hospital stay length.

DETAILED DESCRIPTION:
Discectomy is the most common surgical technique to solve lumbar radiculopathy caused by disc herniation and nerve roots compression .

Currently, microscopic discectomy is performed as a minimally invasive surgery, thus reducing the impact of so-called conventional "open" discectomies.

Minimally invasive spinal surgery was developed using a retractor tube, a microscope, and an endoscope to perform efficient nerves decompression while preserving spinal cord stabilizing structures.

Although more technically demanding, discectomy with full endoscopy made possible a significant reduction of surgery invasive impact, thus making possible to broaden the field of endoscopic surgery indications.

This study is based on hypothesis that full endoscopic discectomy offers several advantages over traditional microscopic discectomy, including a smaller skin incision and therefore fewer scars and less muscle damage, lower infection rate, less blood loss, less painful post-operative recovery and shorter hospital stay length.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient operated under endoscopy for lumbar disc herniation between February 2020 and May 2022
* Patient operated by conventional microscopic surgery for lumbar disc herniation before February 2020
* Patient having been informed of the research and not opposing its data use as part of this research

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need discetomy for lumbar disc herniation
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate within 3 months after discectomy | 3 months
  Number of patients hospitalized within 3 months after surgery will be used to define re hospitalization percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, Toutes, France

IPD SHARING:
Plan to Share IPD: No